CLINICAL TRIAL: NCT02701777
Title: Maximizing Spike - Timing Dependent Plasticity After Spinal Cord Injury
Brief Title: Enhancing STDP After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B1807-R
Record Dates: First submitted 2016-01-14; First posted 2016-03-08 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Spinal Cord Injury
Keywords: spike timing dependant plasticity
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants will not know if they receive real or sham stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- STDP (Active Comparator): Paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  Interventions: Other: STDP
- STDP + Training (Active Comparator): Paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time. Motor training will follow paired stimulation.
  Interventions: Other: STDP; Behavioral: Training
- Sham STDP + Training (Active Comparator): Sham or fake paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined times. Motor training will follow stimulation.
  Interventions: Behavioral: Training; Other: Sham STDP
- Multisite-STDP + Training (Other): Prospective Single Cohort Multisite-Paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time. Motor training will follow paired stimulation.
  Interventions: Behavioral: Training; Other: Multisite-STDP

INTERVENTIONS:
Other: STDP — Paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  Other Names: Paired stimulation
  Arms: STDP; STDP + Training
Behavioral: Training — The participant will be asked to perform exercises using their hands and arms.
  Arms: Multisite-STDP + Training; STDP + Training; Sham STDP + Training
Other: Sham STDP — Sham or fake paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined times.
  Arms: Sham STDP + Training
Other: Multisite-STDP — Paired stimulation will be given to the brain bilaterally, thoracic spine, and several peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  Arms: Multisite-STDP + Training

SUMMARY:
The overall goal is to develop new clinical approaches to restore limb function after spinal cord injury (SCI). Corticospinal tract (CST) axons are involved in controlling limb function. Paired pulse induced spike-timing dependent plasticity (STDP) enhances synaptic strength between residual CST axons and spinal motoneurons (SMNs) resulting in temporary improvements in limb function in humans with incomplete SCI. Motor training will be combined with paired-pulse STDP stimulation to further enhance plasticity and behavioral recovery.

DETAILED DESCRIPTION:
To induce STDP with paired pulse, corticospinal volleys evoked by either transcranial magnetic stimulation over the primary motor cortex for upper extremities or electrical stimulation over the thoracic spine for lower extremities arrive at corticospinal-motor neuronal synapses of upper- or lower-limb muscles, 1-2 ms before antidromic potentials were elicited in motor neurons by electrical stimulation of corresponding peripheral nerves.

ELIGIBILITY:
Inclusion Criteria:

Participants who are unimpaired healthy controls:

* Male and females between ages 18-85 years
* Right handed
* Able to complete precision grips with both hands
* Able to complete full wrist flexion-extension bilaterally
* Able to walk unassisted
* Able to complete full ankle flexion-extension bilaterally

Participants who have had a spinal cord injury:

* Male and females between ages 18-85 years
* SCI ( 6 months of injury)
* Spinal Cord injury at or above L5
* The ability to produce a visible precision grip force with one hand
* Able to perform some small wrist flexion and extension
* The ability to perform a small visible contraction with dorsiflexion and hip flexor muscles
* No subjects will be excluded based on their race, religion, ethnicity, gender or HIV status.
* ASIA A,B,C, or D

Exclusion Criteria:

Exclusion criteria for enrollment For SCI and Healthy Control Subjects (4-8 exclusion for non-invasive brain stimulation only):

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold (see appendix 2)
* Pregnant females
* Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida, MS, or herniated disk
* Individuals with scalp shrapnel, cochlear implants, or aneurysm clips.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Oudega, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- STDP: Paired stimulation (STDP) will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  STDP: Paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  Participants will complete 10 STDP study visits each lasting ~2 hours.
  Baseline and post 10 measurements will be collected for the following measurements:
  Changes in TMS measurements in the form of motor evoked potentials (MEPs). Changes in the maximum voluntary contraction (MVC) will be measured using surface EMG.
  Functional measurements: GRASSP, will measure changes in the time it takes to complete hand tasks; 10-m walk test, will measure changes in walking speed.
  Follow-up measurements will be done after 6 months with available participants for MEPs, MVC, and functional measurements.
- STDP + Training: Paired stimulation (STDP) will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  STDP: Paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  Training: The participant will be asked to perform exercises using their upper and lower extremities.
  Participants will complete 10 STDP + Training study visits each lasting ~2 hours.
  Baseline and post 10 measurements will be collected for the following measurements:
  Changes in TMS measurements in the form of motor evoked potentials (MEPs). Changes in the maximum voluntary contraction (MVC) will be measured using surface EMG.
  Functional measurements: GRASSP, will measure changes in the time it takes to complete hand tasks; 10-m walk test, will measure changes in walking speed.
  Follow-up measurements will be done after 6 months with available participants for MEPs, MVC, and functional measurements.
- Sham STDP + Training: Sham or fake paired stimulation (Sham STDP) will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined times. Motor training will follow stimulation.
  Training: The participant will be asked to perform exercises using their upper and lower extremities.
  Sham STDP: Sham or fake paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined times.
  Participants will complete 10 Sham STDP + Training study visits each lasting ~2 hours.
  Baseline and post 10 measurements will be collected for the following measurements:
  Changes in TMS measurements in the form of motor evoked potentials (MEPs). Changes in the maximum voluntary contraction (MVC) will be measured using surface EMG.
  Functional measurements: GRASSP, will measure changes in the time it takes to complete hand tasks; 10-m walk test, will measure changes in walking speed.
  Follow-up measurements will be done after 6 months with available participants for MEPs, MVC, and functional measurements.
- Multisite-STDP + Training: Prospective Single Cohort Multisite-Paired stimulation (Multisite-STDP) will be given to the brain, spinal cord and peripheral nerves so that the messages are received at the spinal cord at predetermined time. Motor training will follow paired stimulation.
  Multisite-STDP: Paired stimulation will be given to the brain, spinal cord and peripheral nerves so that the messages are received at the spinal cord at predetermined time.
  Training: The participant will be asked to perform exercises using their upper and lower extremities.
  Participants will complete 40 multisite-STDP + Training study visits each lasting ~2 hours.
  Baseline, post 20, and post 40 measurements will be collected for the following measurements:
  Changes in TMS measurements in the form of motor evoked potentials (MEPs). Changes in the maximum voluntary contraction (MVC) will be measured using surface EMG.
  Functional measurements: GRASSP, will measure changes in the time it takes to complete hand tasks; 10-m walk test, will measure changes in walking speed.
  Baseline and post 40 measurements will be collected for the following measurements:
  ISNCSCI, will measure neurologic and functional recovery; SCI-QOL, will measure changes in quality of life functions.
  Follow-up measurements will be done after 9 months with available participants for GRASSP, 10-m walk test, and SCI-QOL.
Period: Overall Study
Arm/Group | STDP | STDP + Training | Sham STDP + Training | Multisite-STDP + Training
Started | 17 | 16 | 16 | 13
Completed | 13 | 13 | 12 | 11
Not Completed | 4 | 3 | 4 | 2
Not completed — Some subjects did not like the stimulation. | 4 | 0 | 0 | 2
Not completed — Some subjects were unable to commit to the training study. | 0 | 3 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STDP | STDP + Training | Sham STDP + Training | Multisite-STDP + Training | Total
Number analyzed (Participants) | 13 | 13 | 12 | 11 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 12 | 8 | 43
  >=65 years | 1 | 2 | 0 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 45.1 [21 to 71] | 45.6 [23 to 82] | 41.8 [22 to 59] | 48.2 [21 to 84] | 45 [21 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 1 | 5 | 14
  Male | 9 | 9 | 11 | 6 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 6 | 2 | 22
  Not Hispanic or Latino | 7 | 5 | 6 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3 | 0 | 6
  Black or African American | 3 | 0 | 5 | 2 | 10
  White | 5 | 5 | 0 | 8 | 18
  More than one race | 5 | 5 | 4 | 1 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 12 | 11 | 49
Time post injury [Mean (Standard Deviation); unit: years] | 7.1 (5.4) | 12.7 (12.5) | 9.1 (6.1) | 8.9 (10.6) | 9.5 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment
Description: The Graded Redefined Assessment of Strength Sensibility and Prehension (GRASSP) assessment is a standardized test of functional abilities of the hand. We measure time required to complete the GRASSP test for upper extremity functional assessment. 10-m walk test is used to measure walking speed for lower extremity functional assessment. The time to complete the task is assessed in seconds for both measurements and normalized as percentage of Baseline. Normalization to baseline allows comparison across two different tasks.
  For STDP, STDP+Training, and Sham-STDP+Training groups, either GRASSP or 10-m walk test was performed in each participant depending on the targeted muscle. For Multisite-STDP + Training group, both GRASSP and 10-m walk test were performed in each participant and the average of two tests were reported below.
Time Frame: Measured at baseline, after 10-20 sessions, and follow up (after 6 months) for STDP, STDP+Training, and Sham-STDP+Training groups . Measured at baseline, after 20 and 40 sessions, and follow up (after 9 months) for Multisite-STDP + Training group.
Population: The number of participants analyzed is different from overall number of participants because some participants could not perform the GRASSP and/or 10-m walk test. Follow-up was performed only with available participants.
Measure: Mean (Standard Deviation); unit: percentage of Baseline
Groups:
- STDP: Paired stimulation (STDP) will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  STDP: Paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  Participants will complete study visits each lasting ~2. Changes in TMS measurements in the form of motor evoked potentials (MEPs) will be measured before and after the 30 minute STDP intervention. The maximum voluntary contraction (MVC) will be measured using surface EMG before and after the 30 minute STDP intervention.
- STDP + Training: Paired stimulation (STDP) will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time. Motor training will follow paired stimulation.
  STDP: Paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined time.
  Training: The participant will be asked to perform exercises using their hands and arms.
  Participants will complete 10 STDP + Training study visits each lasting ~2. Baseline and post measurements will be collected.
  The following measurements were collected:
  Changes in TMS measurements in the form of motor evoked potentials (MEPs). Changes in the maximum voluntary contraction (MVC) will be measured using surface EMG.
  Functional measurement, GRASSP, will measure changes in the time it takes to complete hand tasks.
- Sham STDP + Training: Sham or fake paired stimulation (Sham STDP) will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined times. Motor training will follow stimulation.
  Training: The participant will be asked to perform exercises using their hands and arms.
  Sham STDP: Sham or fake paired stimulation will be given to the brain and to a peripheral nerve so that the messages are received at the spinal cord at predetermined times.
  Participants will complete 10 Sham STDP + Training study visits each lasting ~2.
  Baseline and post measurements will be collected.
  The following measurements were collected:
  Changes in TMS measurements in the form of motor evoked potentials (MEPs). Changes in the maximum voluntary contraction (MVC) will be measured using surface EMG.
  Functional measurement, GRASSP, will measure changes in the time it takes to complete hand tasks.
Arm/Group | STDP | STDP + Training | Sham STDP + Training | Multisite-STDP + Training
Number analyzed (Participants) | 8 | 6 | 8 | 11
percentage of Baseline
  Baseline | 100 (0) | 100 (0) | 100 (0) | 100 (0)
  After 10 sessions: number analyzed (Participants) | 8 | 6 | 8 | 0
  After 10 sessions | 80.5 (9.1) | 75.6 (18.6) | 82.6 (20.1) |
  After 20 sessions: number analyzed (Participants) | 0 | 0 | 0 | 11
  After 20 sessions |  |  |  | 62.4 (10.9)
  After 40 sessions: number analyzed (Participants) | 0 | 0 | 0 | 11
  After 40 sessions |  |  |  | 49.1 (10.9)
  Follow-up: number analyzed (Participants) | 0 | 4 | 5 | 8
  Follow-up |  | 78.4 (9.6) | 100.6 (10.5) | 48.3 (16.5)

2. Secondary Outcome: Amplitude of Motor Evoked Potential (MEP)
Description: We measure amplitude of a motor evoked potential evoked by transcranial magnetic stimulation (TMS) or thoracic spine stimulation. The amplitude of MEP is assessed in millivolts and normalized as percentage of Baseline. Normalization to baseline is necessary to allow comparison across different muscles because the targeted muscle is different for each individual depending on the level of injury.
Time Frame: Measured at baseline, after 10-20 sessions, and follow up (after 6 months) for STDP, STDP+Training, and Sham-STDP+Training groups . Measured at baseline and after 20 and 40 sessions for Multisite-STDP + Training group.
Population: Follow up was done with available participants.
Measure: Mean (Standard Deviation); unit: percentage of Baseline
Arm/Group | STDP | STDP + Training | Sham STDP + Training | Multisite-STDP + Training
Number analyzed (Participants) | 13 | 13 | 12 | 11
percentage of Baseline
  Baseline | 100 (0) | 100 (0) | 100 (0) | 100 (0)
  After 10 sessions: number analyzed (Participants) | 13 | 13 | 12 | 0
  After 10 sessions | 153.2 (40.7) | 164.6 (64.0) | 99.1 (12.4) |
  After 20 sessions: number analyzed (Participants) | 0 | 0 | 0 | 11
  After 20 sessions |  |  |  | 233.2 (65.9)
  After 40 sessions: number analyzed (Participants) | 0 | 0 | 0 | 11
  After 40 sessions |  |  |  | 368.9 (108.9)
  Follow-up: number analyzed (Participants) | 0 | 5 | 5 | 0
  Follow-up |  | 172 (57.7) | 89.0 (22.1) |

3. Secondary Outcome: Maximum Voluntary Contraction
Description: We measure maximum voluntary contraction (MVC) of muscles recorded by electromyography (EMG) in the targeted muscle(s). Average of muscles was reported for Multisite-STDP + Training group. The maximum voluntary contraction is assessed in millivolts and normalized as percentage of Baseline. Normalization to baseline is needed to allow comparison across different muscles because the targeted muscle is different for each individual depending on the level of injury.
Time Frame: as for outcome 2
Population: Follow-up was done only with available participants.
Measure: Mean (Standard Deviation); unit: percentage of Baseline
Arm/Group | STDP | STDP + Training | Sham STDP + Training | Multisite-STDP + Training
Number analyzed (Participants) | 13 | 13 | 12 | 11
percentage of Baseline
  Baseline | 100 (0) | 100 (0) | 100 (0) | 100 (0)
  After 10 sessions: number analyzed (Participants) | 13 | 13 | 12 | 0
  After 10 sessions | 139.4 (23.3) | 144.6 (50.7) | 100.7 (12.3) |
  After 20 sessions: number analyzed (Participants) | 0 | 0 | 0 | 11
  After 20 sessions |  |  |  | 161.0 (49.5)
  After 40 sessions: number analyzed (Participants) | 0 | 0 | 0 | 11
  After 40 sessions |  |  |  | 193.1 (71.0)
  follow-up: number analyzed (Participants) | 0 | 5 | 5 | 0
  follow-up |  | 154.5 (25.0) | 108.8 (7.8) |

4. Secondary Outcome: ISNCSCI-motor Scores
Description: Neurological recovery was measured by the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. Motor part of the exam is completed through the testing of key muscle functions corresponding to 10 myotomes (C5-T1 and L2-S1) for right and left side separately. The strength of each muscle function is graded on a six-point scale ranging from 0 meaning complete paralysis to 5 meaning full strength. The total motor score is sum of all motor scores across 10 myotomes for both sides and therefore ranges from 0-100. Higher scores represent better outcome. We reported the total motor score.
Time Frame: ISNCSCI was performed at baseline and after 40 sessions of Multisite-STDP+Training.
Population: We performed ISNCSCI exam only for "Multiside-STDP+training" group but not in the other groups ("STDP", "STDP + Training" and "Sham STDP + Training"). Therefore the results were provided only for "Multiside-STDP+training" group.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Multisite-STDP + Training
Number analyzed (Participants) | 11
scores on a scale
  Baseline | 59.4 (23.7)
  After 40 sessions | 68.9 (20.2)

5. Secondary Outcome: ISNCSCI-sensory Scores
Description: Neurological recovery was measured by the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. Sensory part of the exam is completed through the testing of a key point in each of the 28 dermatomes (from C2 to S4-5) on the right and left sides of the body. At each of these key points, two aspects of sensation are examined: light touch and pin prick (sharp-dull discrimination). Appreciation of light touch and pin prick sensation at each of the key points is separately scored on a three-point scale; 0-absent, 1-altered, and 2-normal or intact. Therefore, 56 is the maximum score for both light touch and pin prick and the total sensory score ranges from 0 to 112. Higher scores represent better outcome. We reported the total sensory score.
Time Frame: ISNCSCI was performed at baseline and after 40 sessions of Multisite-STDP+Training.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Multisite-STDP + Training
Number analyzed (Participants) | 11
scores on a scale
  Baseline | 99.0 (34.6)
  After 40 sessions | 119.9 (38.4)

6. Secondary Outcome: SCI-QOL-ambulation
Description: We used questionnaire to assess changes in quality of life. The name of the questionnaire is Spinal Cord Injury Quality of Life (SCI-QOL) and we used four subdomains: ambulation, self-care, bowel management difficulties, and bladder management difficulties. Scores on all subdomains of SCI-QOL use a standardized T metric, with a mean of 50 and a standard deviation of 10. Ambulation subdomain assesses the ability to engage in walking activities in different locations that vary based on speed, time and condition and the ability to manage stairs under different conditions. Higher scores on Ambulation subdomain represent better outcome.
Time Frame: Measured at baseline, after 40 sessions, and follow up (after 9 months) for Multisite-STDP + Training group.
Population: We performed SCI-QOL exam only for "Multiside-STDP+training" group but not in the other groups ("STDP", "STDP + Training" and "Sham STDP + Training"). Therefore the results were provided only for "Multiside-STDP+training" group. Follow up was done with available participants.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Multisite-STDP + Training
Number analyzed (Participants) | 11
T-scores
  Baseline | 53.7 (9.4)
  After 40 sessions | 57.1 (7.9)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 61.4 (5.3)

7. Secondary Outcome: SCI-QOL-self-care
Description: We used questionnaire to assess changes in quality of life. The name of the questionnaire is Spinal Cord Injury Quality of Life (SCI-QOL) and we used four subdomains: ambulation, self-care, bowel management difficulties, and bladder management difficulties. Scores on all subdomains of SCI-QOL use a standardized T metric, with a mean of 50 and a standard deviation of 10. Self-care subdomain assesses an individual's ability to perform daily self-care activities such as eating, dressing, grooming, and bathing. Higher scores on Self-care subdomain represent better outcome.
Time Frame: Measured at baseline, after 40 sessions, and follow up (after 9 months) for Multisite-STDP + Training group.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Multisite-STDP + Training
Number analyzed (Participants) | 11
T-scores
  Baseline | 45.9 (7.8)
  After 40 sessions | 47.5 (8.0)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 48.5 (3.6)

8. Secondary Outcome: SCI-QOL- Bowel Management Difficulties
Description: We used questionnaire to assess changes in quality of life. The name of the questionnaire is Spinal Cord Injury Quality of Life (SCI-QOL) and we used four subdomains: ambulation, self-care, bowel management difficulties, and bladder management difficulties. Scores on all subdomains of SCI-QOL use a standardized T metric, with a mean of 50 and a standard deviation of 10. Bowel management difficulties subdomain measures a range of difficulties associated with bowel management, including an ability to carry out a bowel program; concerns about incontinence and bowel accidents; concerns about difficulty implementing a bowel program; and the impact of bowel management on everyday living. Higher scores on bowel management difficulties subdomain represent better outcome.
Time Frame: Measured at baseline, after 40 sessions, and follow up (after 9 months) for Multisite-STDP + Training group.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Multisite-STDP + Training
Number analyzed (Participants) | 11
T-scores
  Baseline | 48.2 (10.6)
  After 40 sessions | 51.8 (10.7)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 45.4 (7.3)

9. Secondary Outcome: SCI-QOL- Bladder Management Difficulties
Description: We used questionnaire to assess changes in quality of life. The name of the questionnaire is Spinal Cord Injury Quality of Life (SCI-QOL) and we used four subdomains: ambulation, self-care, bowel management difficulties, and bladder management difficulties. Scores on all subdomains of SCI-QOL use a standardized T metric, with a mean of 50 and a standard deviation of 10. Bladder management difficulties subdomain measures a range of difficulties associated with bladder management, including ability to carry out a bladder program; worry about bladder accidents; concerns about implementing one's bladder program; and impact on everyday living. Higher scores on bladder management difficulties subdomain represent better outcome.
Time Frame: Measured at baseline, after 40 sessions, and follow up (after 9 months) for Multisite-STDP + Training group.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Multisite-STDP + Training
Number analyzed (Participants) | 11
T-scores
  Baseline | 41.0 (9.5)
  After 40 sessions | 46.7 (7.6)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 40.9 (7.6)

ADVERSE EVENTS:
Time Frame: The adverse event data is collected from baseline to completion of study visits, an average of 2~3 weeks for Arms 1-3. The longer experiment, Arm 4, involves ~50 visits (40 sessions + baseline, post 20, post 40, and follow-up assessments). This gives a total of 10~15 weeks.
Description: Arm 1 includes all participants who were monitored for adverse events even if they did not complete the study visit.
Arm/Group | STDP | STDP + Training | Sham STDP + Training | Multisite-STDP + Training
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/16 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT02701777/Prot_SAP_001.pdf